CLINICAL TRIAL: NCT02402621
Title: Comparison Between Conventional and Model-based Infusion Strategy of Intravenous Patient-controlled Analgesia in Patients Undergoing Robot Assisted Laparoscopic Radical Prostatectomy
Brief Title: Comparison Between Conventional and Model-based Infusion Strategy of IV PCA in Patients Undergoing RALP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Asan Medical Center (Other)
Responsible Party: Principal Investigator, Young-Kug Kim, Professor, Asan Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2015-0267
Record Dates: First submitted 2015-03-23; First posted 2015-03-30 (Estimated); Last update posted 2015-12-02 (Estimated); Status verified 2015-11

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Fentanyl

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Conventional analgesic group (Active Comparator): fentanyl
  Interventions: Drug: fentanyl
- Model based analgesic group (Experimental): fentanyl
  Interventions: Drug: fentanyl

INTERVENTIONS:
Drug: fentanyl — fentanyl with antiemetic drug

SUMMARY:
Comparing postoperative analgesics requirements and complications between conventional and model-based infusion strategy of intravenous patient-controlled analgesia in patients who undergoing robot assisted laparoscopic radical prostatectomy

Group A: conventional intravenous patient-controlled analgesia, Group B: model-based infusion strategy of intravenous patient-controlled analgesia

DETAILED DESCRIPTION:
The investigators compared postoperative analgesics requirements and complications between conventional and model-based infusion strategy of intravenous patient-controlled analgesia (IV PCA) in patients who undergoing robot assisted laparoscopic radical prostatectomy (RALP)

Group A: conventional IV PCA, Group B: model based IV PCA

1. Primary endpoint: comparison of postoperative analgesic requirements in patient undergoing robot assisted laparoscopic radical prostatectomy (RALP) between conventional patient controlled analgesia (PCA) (Group A) and effective-compartment based dosing strategy of PCA (Group B)
2. Secondary endpoint: 1) VAS analysis between two groups, 2) postoperative nausea and vomiting analysis between two groups, 3) complication evaluation between two groups

ELIGIBILITY:
Inclusion Criteria:

* Patient who is scheduled to get a robot assisted laparoscopic radical prostatectomy
* Patient who agree to get a patient controlled analgesia

Exclusion Criteria:

* American Society of Anesthesiologist (ASA) physical status over III
* History of alcohol or drug addiction
* History of acute or chronic pain or pain treatment
* Allergic to opioid analgesics
* BMI over 30 kg/m2
* History of sleep apnea or respiratory complications

Ages: 20 Years to 69 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 111 (Actual)
Dates: Start 2015-04; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Amount and number of postoperative analgesic requirements | Participants will be followed for the duration of hospital stay, an expected average of 1 week

SECONDARY OUTCOMES:
Number of participants with complications | Up to 48 hours
Visual Analog Scale (VAS) | Up to 48 hours
Postoperative nausea and vomiting | Up to 48 hours
Respiratory rate, oxygen saturation | Up to 48 hours

CONTACTS AND LOCATIONS:
Overall Officials: Young-Kug Kim, Principal Investigator — Asan Medical Center
Locations (1):
- Asan Medical Center, Seoul, South Korea